CLINICAL TRIAL: NCT04330287
Title: A Prospective, Epidemiologic and Multicentre Trial to Determine the Cardiovascular Risk, New Cardiovascular Events and the Cardiovascular Diseases in HIV-infected Patients: 15 Year Follow up
Brief Title: HIV-HEART Aging Study
Acronym: HIVH
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Stefan Esser M.D., Prof. M.D. Head of HPSTD Ambulance, University Hospital, Essen, Principal Investigator, University Hospital, Essen
Other Study IDs: 14-5874-BO
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: HIV Infections; Coronary Disease; Myocardial Infarction; HIV Encephalopathy; Aging; Heart Failure; Weight Gain
Keywords: HIV; AIDS; Antiretroviral therapy; Aging; Heart Failure; coronary heart desease; myocardial infarction; HIV-associated neurocognitive disorders; weight gain
MeSH Terms: conditions — HIV Infections; Coronary Disease; Myocardial Infarction; AIDS Dementia Complex; Heart Failure; Weight Gain; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — stored blood and stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The HIV/HEART Aging study (HIVH) is an ongoing, prospective, multicentre trial that was conducted to assess the incidence, the prevalence and the clinical course of cardiovascular diseases (CVD) in HIV-infected patients. The study population includes outpatients from specialized HIV-care units of the German Ruhr region, who were at least 18 years of age, were known to have a HIV-infection and exhibited a stable disease status within 4 weeks before inclusion into the trial. From March 2004 (Pilot phase) to October 2022 (15 year Follow-up) 1858 HIV+ patients were recruited in a consecutive manner. The standardised examinations included a targeted assessment of medical history and physical examination. Blood was drawn for comprehensive laboratory tests including HIV specific parameters (CD4 cell count, HIV-1 RNA levels) and cardiovascular items (lipid concentrations, BNP values and renal parameters). Furthermore, non-invasive tests were performed during the initial visit, including additional heart rate and blood pressure measurements, electrocardiogram (ECGs) and transthoracic echocardiography (TTE). Examinations were completed in accordance with previously defined standard operating procedures. CVD were defined as coronary, cerebrovascular, peripheral arterial disease, heart failure or cardiac vitium.

DETAILED DESCRIPTION:
A comprehensive detailed description of the study procedures had been previously published (European Journal of medical research 2007;12:243-248).

Comprehensive non invasive cardiovascular examination

* Anamnesis
* File recherche,Physical examination
* Documentation of the cardiovascular and antiretroviral medical therapy
* Electrocardiogram
* Transthoracic echocardiography (optional)
* Exercise electrocardiogram (optional)
* Exercise Montreal Cognitive Assessment test (optional)
* Exercise the Grooved Pegboard test (optional)
* Blood and stool sample collection (optional)
* Questionnaire to quality of life and health economics

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Known HIV-infection
* Signed informed consent

Exclusion Criteria:

* Acute cardiovascular disease
* Unstable hemodynamic status in the three weeks before inclusion
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: population affected by HIV
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-05-11 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of frequency, severity of cardiovascular diseases - especially of coronary artery disease - in patients with HIV-Infection | Baseline up to 15 year follow up
  Calculation of the Framingham Risk Score. It was assumed, that in the next 10 years the individual cardiovascular risk varies between maximal 20% and minimal 0%.
Detection of progression of cardiovascular diseases - especially of coronary artery disease - in patients with HIV-Infection | Baseline up to 15 year follow up
  Calculation of Odds Ratio

SECONDARY OUTCOMES:
Impact on cardiovascular risk on amount of atherosclerosis | Baseline up to 15 year follow up
  in relation to age, gender and classic cardiovascular rsik factors inter alia smoking, diabetes, hypercholesterinaemia and arterial hypertension by calculating the relative risk
Impact on life quality | Baseline up to 15 year follow up
  in relation to HIV-specfic cardiovascular rsik factors including inter alia virus load (copies/ml) in combination with CD4-count and duration of HV-Infection by calculating the standard deviation
Impact on life quality | Baseline up to 15 year follow up
  in relation to HIV-specfic cardiovascular rsik factors including inter alia CD4-count (cells/mm3) in combination with virus load and duration of HIV-infection by calculating the standard deviation
Impact on life quality | Baseline up to 15 year follow up
  in relation to HIV-specfic cardiovascular rsik factors including inter alia duration of HIV-Infection (in years) in combination with virus load and CD4-count by calculating the standard deviation
Impact on cardiovascular risk, amount of atherosclerosis and life quality | Baseline up to 15 year follow up
  in relation to cardiovascular and antiretroviral medication by calculating the 95%-Confidence interval

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - Universitätsklinikum Essen, Klinik für Dermatologie, Essen, Nordrheinwestfalen
  - HIV physician pratice, Duisburg, North Rhine-Westphalia
  - Institut für Medizinische Informatik, Biometrie und Epidemiologie, Essen, North Rhine-Westphalia
  - University Hospital of Bochum, Department of Dermatology, Bochum
  - HIV Outpatient Department, Dortmund

REFERENCES:
- [Result] Kehrmann J, Menzel J, Saeedghalati M, Obeid R, Schulze C, Holzendorf V, Farahpour F, Reinsch N, Klein-Hitpass L, Streeck H, Hoffmann D, Buer J, Esser S; HIV-HEART Study Group. Gut Microbiota in Human Immunodeficiency Virus-Infected Individuals Linked to Coronary Heart Disease. J Infect Dis. 2019 Jan 9;219(3):497-508. doi: 10.1093/infdis/jiy524. PMID 30202890
- [Result] Reinsch N, Streeck H, Holzendorf V, Schulze C, Neumann T, Brockmeyer NH, Kehrmann J, Schadendorf D, Esser S; HIV HEART Study Group. B-type natriuretic peptides for the prediction of cardiovascular events and mortality in patients living with HIV: Results from the HIV-HEART study. Int J Cardiol. 2019 Apr 15;281:127-132. doi: 10.1016/j.ijcard.2019.01.066. Epub 2019 Jan 23. PMID 30711264
- [Result] Schulz CA, Mavarani L, Reinsch N, Albayrak-Rena S, Potthoff A, Brockmeyer N, Hower M, Erbel R, Jockel KH, Schmidt B, Esser S; HIV HEART Aging Study Group and Heinz Nixdorf Recall Investigative Group. Prediction of future cardiovascular events by Framingham, SCORE and asCVD risk scores is less accurate in HIV-positive individuals from the HIV-HEART Study compared with the general population. HIV Med. 2021 Sep;22(8):732-741. doi: 10.1111/hiv.13124. Epub 2021 May 24. PMID 34028959
- [Result] Mavarani L, Albayrak-Rena S, Potthoff A, Hower M, Dolff S, Sammet S, Maischack F, Schadendorf D, Schmidt B, Esser S; HIV HEART AGING Study. Changes in body mass index, weight, and waist-to-hip ratio over five years in HIV-positive individuals in the HIV Heart Aging Study compared to the general population. Infection. 2023 Aug;51(4):1081-1091. doi: 10.1007/s15010-023-02009-8. Epub 2023 Mar 17. PMID 36930373
- [Derived] Mavarani L, Reinsch N, Albayrak-Rena S, Potthoff A, Hower M, Dolff S, Schadendorf D, Jockel KH, Schmidt B, Esser S. The Association of HIV-Specific Risk Factors with Cardiovascular Events in Addition to Traditional Risk Factors in People Living with HIV. AIDS Res Hum Retroviruses. 2024 Apr;40(4):235-245. doi: 10.1089/AID.2023.0055. Epub 2023 Oct 9. PMID 37675901